CLINICAL TRIAL: NCT00092924
Title: A Phase 2, Multi-Center, Open-Label Study to Evaluate the Efficacy, Safety, and Tolerability of TRM-1 (Fully Human Monoclonal Antibody To TRAIL-R1) in Subjects With Relapsed or Refractory Non-Small Cell Lung Cancer
Brief Title: Study of TRM-1(TRAIL-R1 Monoclonal Antibody) in Subjects With Relapsed or Refractory Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRM1-ST03
Record Dates: First submitted 2004-09-24; First posted 2004-09-28 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — mapatumumab

INTERVENTIONS:
Drug: TRAIL-R1 mAb (TRM-1;HGS-ETR1)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TRM-1 in subjects with relapsed or refractory non-small cell lung cancer.

ELIGIBILITY:
Primary Inclusion Criteria:

* Relapsed or refractory histologically or cytologically confirmed Stage IIIB, IV, or recurrent NSCLC
* Previously treated and failed to respond to standard therapy or progressed after standard therapy
* 18 years of age or older

Primary Exclusion Criteria:

* Received a non-FDA approved investigational agent within the last 4 weeks.
* Previous cancer therapies (chemotherapy, hormonal therapy, monoclonal antibodies or radiation therapy) within the last 3 weeks, 8 weeks for fully human or humanized monoclonal antibodies
* Infection requiring antibiotics or hospitalization within the last 2 weeks
* HIV, Hepatitis-B, Hepatitis-C
* Pregnant or breast-feeding women
* Major surgery within the last 4 weeks
* History of other cancers within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2005-01 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (5):
  - University of Colorado Cancer Center, Denver, Colorado
  - Rush Medical College, Chicago, Illinois
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - MD Anderson, Houston, Texas